CLINICAL TRIAL: NCT04214041
Title: Soft Tissue Volume Augmentation of Localized Horizontal Ridge Defects Using Autologous Fat Grafting Versus Subepithelial Connective Tissue Graft (a Randomized Controlled Clinical Trial)
Brief Title: Autologous Fat Grafting Versus Subepithelial Connective Tissue Graft for Volume Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Instructor of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: fat vs subepithelial CT graft
Record Dates: First submitted 2019-12-26; First posted 2019-12-30 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: This non-inferiority study was designed as a randomized controlled clinical trial including 26 localized horizontal ridge defects that were equally allocated (1:1) into one of two parallel groups.
Who Masked: Outcomes Assessor
Masking Description: Neither the operator nor the participants could be blinded to the treatment type as the intervention procedures were markedly different between test and control groups. To enable blinding during outcome assessment, the stereolithography (STL) files of digitized casts were given a code different from that of the allocation procedure and were kept confidential. The volumetric analysis was performed and the groupings were shared with the biostatistician as groups A and B. Only during the interpretation the codes and groups were translated into test and control groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous fat grafting (Experimental)
  Interventions: Other: Autologous fat grafting
- Sub-epithelial connective tissue graft (Active Comparator)
  Interventions: Other: Sub-epithelial connective tissue graft

INTERVENTIONS:
Other: Autologous fat grafting — A fat graft will be aspirated from the abdomen under local anaesthesia and processed using the Microfat grafting technique. Afterwards the fat graft will be injected in the previously created pouch at the recipient site. Then the pouch will be closed using interrupted sutures 5-0 vicryl.
  Arms: Autologous fat grafting
Other: Sub-epithelial connective tissue graft — A subepithelial connective tissue graft of a size that corresponds to that of the defect will be harvested from the palate using the trap door technique. The donor site will be closed using cross horizontal sling sutures and interrupted sutures 4-0 vicryl. Subsequently, the graft will be inserted in the previously created pouch at the recipient site and secured to the flap using vicryl sutures 5-0. Then the pouch will be closed using interrupted sutures.
  Arms: Sub-epithelial connective tissue graft

SUMMARY:
The aim of this study was to evaluate the effectiveness of autologous fat as a grafting material for soft tissue volume augmentation of localized horizontal ridge defects in humans.

DETAILED DESCRIPTION:
A total of 20 patients having 26 localized horizontal ridge defects were recruited for the study from the patient pool at the dental clinics of the faculty of dentistry, Alexandria University. Ridge defects were divided into two parallel groups:

Test group: localized ridge defects were augmented using autologous fat grafting Control group: localized ridge defects were augmented using conventional subepithelial connective tissue graft.

ELIGIBILITY:
Inclusion Criteria:

1. Patients had at least one localized horizontal ridge defect in a single tooth gap requiring soft tissue volume augmentation.
2. Teeth in the defect area have been extracted at least 3 months prior to enrolment
3. All patients were systemically healthy
4. Patients were non-smokers
5. Patients had abdominal fat accumulation allowing liposuction
6. Ability to understand the nature of the proposed surgery and ability to sign an informed consent form

Exclusion Criteria:

1. General contra-indications to surgical procedures
2. Pregnancy
3. Systemic diseases like Diabetes Mellitus and autoimmune diseases
4. History of malignancy, chemotherapy or radiotherapy within the last 5 years
5. Concurrent medication affecting mucosal healing in general (e.g. steroids, large doses of anti-inflammatory drugs)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
Volumetric analysis to evaluate soft tissue volume changes | 1 month
  To evaluate the volumetric changes of soft tissues, all the stone models will be digitized using a lab-based optical scanner. The digital surface models will be imported as STL files into the image analysis software for volumetric analysis. Digital cast models representing the different time points during the follow up will be superimposed using tooth surfaces as references. The relevant area for the measurements of volume changes will be defined and volume changes will be calculated by the same examiner according to previous studies
Volumetric analysis to evaluate soft tissue volume changes | 2 months
  To evaluate the volumetric changes of soft tissues, all the stone models will be digitized using a lab-based optical scanner. The digital surface models will be imported as STL files into the image analysis software for volumetric analysis. Digital cast models representing the different time points during the follow up will be superimposed using tooth surfaces as references. The relevant area for the measurements of volume changes will be defined and volume changes will be calculated by the same examiner according to previous studies
Volumetric analysis to evaluate soft tissue volume changes | 3 months
  To evaluate the volumetric changes of soft tissues, all the stone models will be digitized using a lab-based optical scanner. The digital surface models will be imported as STL files into the image analysis software for volumetric analysis. Digital cast models representing the different time points during the follow up will be superimposed using tooth surfaces as references. The relevant area for the measurements of volume changes will be defined and volume changes will be calculated by the same examiner according to previous studies

SECONDARY OUTCOMES:
Probing depth | 1 month
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) at 6 points around the tooth
Probing depth | 2 months
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) at 6 points around the tooth
Probing depth | 3 months
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) at 6 points around the tooth
Clinical attachment loss (CAL) | 1 month
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) at 6 points around the tooth
Clinical attachment loss (CAL) | 2 months
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) at 6 points around the tooth
Clinical attachment loss (CAL) | 3 months
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) at 6 points around the tooth
Bleeding on probing | 1 month
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) and recorded as present/absent
Bleeding on probing | 2 months
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) and recorded as present/absent
Bleeding on probing | 3 months
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) and recorded as present/absent
Width of Keratinized tissue | 1 month
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) and it represents the edentulous span measured at the midpoint between teeth on either side of the edentulous space mesiodistally, starting at the buccal edge of the crest of the ridge till the mucogingival line.
Width of Keratinized tissue | 2 months
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) and it represents the edentulous span measured at the midpoint between teeth on either side of the edentulous space mesiodistally, starting at the buccal edge of the crest of the ridge till the mucogingival line.
Width of Keratinized tissue | 3 months
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) and it represents the edentulous span measured at the midpoint between teeth on either side of the edentulous space mesiodistally, starting at the buccal edge of the crest of the ridge till the mucogingival line.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine Gaweesh, PhD, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Maha A Abou Khadr, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Hussein S Abulhassan, PhD, Study Chair — Faculty of Medicine, Alexandria University, Egypt; Nesma M Khalil, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Del Pizzo M, Modica F, Bethaz N, Priotto P, Romagnoli R. The connective tissue graft: a comparative clinical evaluation of wound healing at the palatal donor site. A preliminary study. J Clin Periodontol. 2002 Sep;29(9):848-54. doi: 10.1034/j.1600-051x.2002.290910.x. PMID 12423299
- [Background] Akcali A, Schneider D, Unlu F, Bicakci N, Kose T, Hammerle CH. Soft tissue augmentation of ridge defects in the maxillary anterior area using two different methods: a randomized controlled clinical trial. Clin Oral Implants Res. 2015 Jun;26(6):688-95. doi: 10.1111/clr.12368. Epub 2014 Apr 10. PMID 24720375
- [Background] Zeltner M, Jung RE, Hammerle CH, Husler J, Thoma DS. Randomized controlled clinical study comparing a volume-stable collagen matrix to autogenous connective tissue grafts for soft tissue augmentation at implant sites: linear volumetric soft tissue changes up to 3 months. J Clin Periodontol. 2017 Apr;44(4):446-453. doi: 10.1111/jcpe.12697. Epub 2017 Feb 11. PMID 28107560
- [Background] Marwah M, Kulkarni A, Godse K, Abhyankar S, Patil S, Nadkarni N. Fat Ful'fill'ment: A Review of Autologous Fat Grafting. J Cutan Aesthet Surg. 2013 Jul;6(3):132-8. doi: 10.4103/0974-2077.118402. PMID 24163528
- [Background] Alharbi Z, Oplander C, Almakadi S, Fritz A, Vogt M, Pallua N. Conventional vs. micro-fat harvesting: how fat harvesting technique affects tissue-engineering approaches using adipose tissue-derived stem/stromal cells. J Plast Reconstr Aesthet Surg. 2013 Sep;66(9):1271-8. doi: 10.1016/j.bjps.2013.04.015. Epub 2013 Jun 2. PMID 23732072
- [Background] Rojo E, Stroppa G, Sanz-Martin I, Gonzalez-Martin O, Alemany AS, Nart J. Soft tissue volume gain around dental implants using autogenous subepithelial connective tissue grafts harvested from the lateral palate or tuberosity area. A randomized controlled clinical study. J Clin Periodontol. 2018 Apr;45(4):495-503. doi: 10.1111/jcpe.12869. Epub 2018 Feb 23. PMID 29334403
- [Background] Schneider D, Ender A, Truninger T, Leutert C, Sahrmann P, Roos M, Schmidlin P. Comparison between clinical and digital soft tissue measurements. J Esthet Restor Dent. 2014 May-Jun;26(3):191-9. doi: 10.1111/jerd.12084. Epub 2013 Dec 17. PMID 24341747
- [Background] Windisch SI, Jung RE, Sailer I, Studer SP, Ender A, Hammerle CH. A new optical method to evaluate three-dimensional volume changes of alveolar contours: a methodological in vitro study. Clin Oral Implants Res. 2007 Oct;18(5):545-51. doi: 10.1111/j.1600-0501.2007.01382.x. Epub 2007 Jun 21. PMID 17590160
- [Background] Fickl S, Schneider D, Zuhr O, Hinze M, Ender A, Jung RE, Hurzeler MB. Dimensional changes of the ridge contour after socket preservation and buccal overbuilding: an animal study. J Clin Periodontol. 2009 May;36(5):442-8. doi: 10.1111/j.1600-051X.2009.01381.x. PMID 19419446